CLINICAL TRIAL: NCT04282291
Title: Serratus Intercostal Plane Block in Supraumbilical Surgery: A Prospective Randomized Comparison
Brief Title: Serratus Intercostal Plane Block,New Analgesia in Supraumbilical Surgery
Acronym: SIPB
Status: Completed | Type: Observational
Sponsor: Hospital Medina del Campo (Other)
Responsible Party: Principal Investigator, María Teresa Fernandez, Principal Investigator, Hospital Medina del Campo
Other Study IDs: PI 16-354
Record Dates: First submitted 2020-02-18; First posted 2020-02-24 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Postoperative Pain; Analgesia; Local Anaesthetic; Abdominal Injury
Keywords: Analgesia; Abdominal surgery
MeSH Terms: conditions — Pain, Postoperative; Agnosia; Abdominal Injuries | interventions — Morphine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 102 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- SIPB (block): patients who underwent a modified BRILMA (intercostal rami block, middle axilary line) ultrasound-guided block with portable device with lineal probe and needle 80 mm. With the patient lying supine, the probe was placed in the sagittal plane of the middle axillary line to identify the aim thoracic structures. Under aseptic conditions, the needle was inserted in plane, caudo-craneal, to reach the fascial plane between the serratus anterior muscle and the external intercostal muscle at the eighth rib. A bolus dose of levobupivacaine 0.25% was administered, 3 ml of local anesthetic for each segment we want to block
  Interventions: Procedure: fascial block as postoperative analgesia; Device: PCA CADD Smith Medical pumps
- control (morphine): PCA (patient controlled analgesia) morphine was initiated immediately postoperatively using CADD Smith Medical pumps. All patients received PCA-morphine with the initial dose being 0.5-1 mg. The bolus dose was 0.01mg/kg mg morphine, with lockout time interval of 15 - 30 min, limiting of 8mg/hour, as the default program. The continuous (basal) dose was increased after 12-24 hours if using frequent demand doses or if pain not controlled and decreasing if no bolus was taken.
  Interventions: Drug: Morphine; Device: PCA CADD Smith Medical pumps

INTERVENTIONS:
Procedure: fascial block as postoperative analgesia — The tissue damage induced by the surgery generates a nociceptive pain which is accompanied by inflammatory mechanism (somatic pain), visceral and neuropathic pain, and why the treatment must be adapted to each surgical procedure. As the innervation of the upper abdominal wall depends mainly on the last intercostal nerves, the block of these nerves should be considered a good analgesic strategy to avoid the somatic pain. The placement of the local anesthetic in the serratus intercostal plane at the eighth rib (serratus intercostal plane block, SIPB) in the middle axillary line, managed to block the lateral and anterior cutaneous branches of the last intercostal nerves (T7-11). The results were satisfactory in the postoperative pain control of the patients with open cholecystectomy.
  Groups: SIPB (block)
Drug: Morphine — The continuous (basal) dose
  Groups: control (morphine)
Device: PCA CADD Smith Medical pumps — perfusion

SUMMARY:
Background: The surgeries with upper abdominal wall incisions cause a severe pain and providing an adequate analgesia is an important challenge for the anesthesiologist. The serratus intercostal plane block (SIPB) has been already described as analgesic technique in open cholecystectomy.

The aim of this study is to evaluate its analgesic efficacy in pain control, opioids consumption and recovery quality in upper abdominal surgeries.

Methods: This blind, randomized controlled study was conducted on 102 patients undergoing open upper abdominal wall surgery under general anesthesia. All patients who received serratus intercostal plane block at the eighth rib as analgesic technique were included in group 0 (SIPB) and in Group 1 (control) those who received continuous intravenous morphine analgesia. In each group was evaluated pain scores in numeric verbal scale (NVS) and opioids consumption at 0,6,12,24 y 48h postoperative time. The quality of the postoperative recovery was evaluated with the modified Postoperative Quality of Recovery Score ( QoR-15 questionnaire) at 24h.

DETAILED DESCRIPTION:
The scientific evidence always supports the employment of a multimodal analgesic strategy, especially in procedures that generate a severe postoperative pain2, as media laparotomy or subcostal incision. The purpose is to not retard the patients' recovery and to avoid complications. The thoracic epidural analgesia is still the reference analgesic technique in open abdominal surgery7, although it is not exempt of limitations and complications. That is why, since the introduction of thoracic and abdominal fascial blocks, they have been part of the analgesic strategy, being an alternative to considerer instead the epidural.

ELIGIBILITY:
Inclusion Criteria:

* informed consent signature
* patients >18 years old,

  . American Society of Anesthesiologist (ASA) risk scale < IV,
* supraumbilical laparotomy (elective laparotomy or laparoscopy conversion)

Exclusion Criteria:

* neurologic impairment,
* inability to give informed consent,
* used drugs allergy,
* contraindications to nerve block (coagulopathy, local infection at the site of the block)
* chronic pain treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: After the informed consent signature the patients were randomly allocated into two groups (1:1 allocation ratio) using a computerized random number generator (http://www.randomization.com). Before the surgery, and with inclusion criteria checked, patients' demographic data were collected (age, sex, ASA risk scale).
Sampling Method: Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2016-02-18 (Actual); Primary Completion 2016-08-01 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
the local anesthetic in the serratus intercostal space at the eighth rib (SIPB)is an opioids sparing method in the perioperative time | 24 postoperative hours
  In a questionnaire designed for the study the pain scores were registered as main outcome, using verbal numeric scale (VNS) from 0(no pain at all) to 10 (worst imaginable pain) both at rest and the dynamic component (cough, deep breath, movement, so on). They were scored at 0, 6,12, 24 and 48 hours postoperatively.

SECONDARY OUTCOMES:
analgesic rescue needed | 48 hours
  intraoperative fentanyl and postoperative morphine
quality of recovery: QoR-15 questionnaire | 24 hours
  using the scale of surgical recovery modified Postoperative Quality of Recovery Score
  (The QoR-15:15 answers) that the patients filled in at 24 hours postoperatively. The QoR-15 questionnaire collected 9 parameters that valued the physical well-being (pain 2 items, Physical Comfort 4 Physical Independence 2) and 6 that valued the mental well-being (Psychological support 2, Emotional state 4). Each scored on an 11 point numerical rating (0-10)

CONTACTS AND LOCATIONS:
Locations (1):
- María Teresa Fernandez, Valladolid, Castille and León, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hamilton DL, Manickam BP. Is a Thoracic Fascial Plane Block the Answer to Upper Abdominal Wall Analgesia? Reg Anesth Pain Med. 2018 Nov;43(8):891-892. doi: 10.1097/AAP.0000000000000838. No abstract available. PMID 30339615
- [Background] Fernandez MT, Lopez S, Ortigosa E. Reply to Dr Wang et al: serratus-intercostal block as opioids-saving strategy in supraumbilical surgery. Reg Anesth Pain Med. 2019 Feb 16:rapm-2019-100384. doi: 10.1136/rapm-2019-100384. Online ahead of print. No abstract available. PMID 30772819
- [Background] Fernandez Martin MT, Lopez Alvarez S, Sanllorente Sebastian R. Serratus anterior plane block for upper abdominal incisions has been previously reported. Anaesth Intensive Care. 2019 Sep;47(5):472-473. doi: 10.1177/0310057X19870546. Epub 2019 Aug 25. No abstract available. PMID 31446767
- [Result] Fernandez Martin MT, Lopez Alvarez S, Mozo Herrera G, Platero Burgos JJ. [Ultrasound-guided cutaneous intercostal branches nerves block: A good analgesic alternative for gallbladder open surgery]. Rev Esp Anestesiol Reanim. 2015 Dec;62(10):580-4. doi: 10.1016/j.redar.2015.02.011. Epub 2015 Apr 17. Spanish. PMID 25896736
- [Result] Fernandez Martin MT, Lopez Alvarez S, Perez Herrero MA. Serratus-intercostal interfascial block as an opioid-saving strategy in supra-umbilical open surgery. Rev Esp Anestesiol Reanim (Engl Ed). 2018 Oct;65(8):456-460. doi: 10.1016/j.redar.2018.03.007. Epub 2018 May 20. English, Spanish. PMID 29789137